CLINICAL TRIAL: NCT01265875
Title: Secretin Infusion for Pain Due to Chronic Pancreatitis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ChiRhoClin, Inc. (Industry)
Collaborators: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-01
Record Dates: First submitted 2010-12-22; First posted 2010-12-23 (Estimated); Results first posted 2016-03-01 (Estimated); Last update posted 2016-03-09 (Estimated); Status verified 2016-03

CONDITIONS: Chronic Pancreatitis
Keywords: Chronic Pancreatitis
MeSH Terms: conditions — Pancreatitis, Chronic | interventions — Secretin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- human secretin (Other): intravenous secretin administration in escalating doses three times daily for three days. After each infusion (1 to 3 hours), at Day 7 after infusion, and at Day 30 after infusion.
  Interventions: Drug: Human Secretin

INTERVENTIONS:
Drug: Human Secretin — Dose Escalation
  Other Names: ChiRhoStim

SUMMARY:
* To determine if intravenous secretin administration in escalating doses three times daily for three days will improve the pain from CP at the time of infusion, after each infusion (1 to 3 hours), at Day 7 after infusion, and at Day 30 after infusion.
* To validate the safety of intravenous secretin administration at the dosage indicated in this study.

DETAILED DESCRIPTION:
12 patients will be enrolled in this study. Patients will be only those treated at Dartmouth-Hitchcock Medical Center for the diagnosis of CP. The diagnosis of CP will be made by the PI based on standard clinical, radiographic and/or biochemical criteria. Patients must be taking prescribed opioid analgesics for the specific treatment of CP at the time of study enrollment. Only patients between the ages of 18-70 and capable of providing informed consent will be considered eligible for the study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, between the ages of 18-70 years old.
2. Documented chronic pancreatitis as determined by CT scan, endoscopic ultrasound, MRCP and/or pancreatic function tests.
3. If female, and not more than 1 year post-menopausal or surgically sterile, must use medically acceptable form of contraception or abstain from sexual activity during the study. Acceptable methods of birth control are: intrauterine device, implantable progesterone device, progesterone intramuscular injection, oral contraceptive (started at least one month prior to Screening Visit 1 and continuing for the duration of the trial), contraceptive patch, condoms with spermicide or abstinence.
4. If a female of reproductive potential, receive counseling on pregnancy protection and effective contraception within 30 days prior to dosing with secretin.
5. Negative serum pregnancy within 72 hours of secretin administration.
6. Use of opioid analgesics for chronic pain from CP.
7. Willing and able to sign written informed consent.

Exclusion Criteria:

1. Male or female <18 or >70 years of age.
2. Abnormal serum amylase and/or lipase indicative of acute pancreatitis within 30 days of study enrollment.
3. Exhibiting signs and/or symptoms of an episode of acute pancreatitis.
4. Severe cardiac disease (stable or unstable angina, congestive heart failure, uncontrolled arrhythmias, implantable defibrillator, severe valvular disease, etc).
5. Severe pulmonary disease (COPD, severe asthma, interstitial lung disease, etc).
6. Severe renal disease (history of acute or chronic renal failure, dialysis dependent, baseline creatinine >2.0 mg/dL).
7. Previous adverse drug event to intravenous secretin.
8. Ongoing illicit drug use or abuse.
9. Ongoing moderate or severe alcohol use defined as greater than 8 oz beer, 8 oz wine and/or 1 oz liquor /day.
10. Acute pancreatitis as defined by the Atlanta Classification definition (refer to Table 1) within the previous two months or symptoms consistent with ongoing acute pancreatitis.
11. Prior pancreatic surgery.
12. Pregnant women, nursing mothers, or women of childbearing potential not employing appropriate contraception.
13. Use of medication that can potentially cause pancreatitis, such as metronidazole, tetracycline, sulfonamides within 30 days prior to Visit 1.
14. Any medical condition which, in the judgment of the investigator, renders participation in this study medically inadvisable.
15. Participation in an investigational clinical study for a drug or medical device within 30 days prior to Visit 1.
16. Unwilling or unable to give written, informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-12; Primary Completion 2011-12 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy B Gardner, M.D., Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire, United States

REFERENCES:
- [Derived] Levenick JM, Andrews CL, Purich ED, Gordon SR, Gardner TB. A phase II trial of human secretin infusion for refractory type B pain in chronic pancreatitis. Pancreas. 2013 May;42(4):596-600. doi: 10.1097/MPA.0b013e318273f3ec. PMID 23548879

RESULTS

PARTICIPANT FLOW:
Groups:
- Human Secretin: Human Secretin : Dose Escalation
  There were 3 days of dosing, 3 doses per day. This was a dose escalation within the participant and did not exceed 0.8mcg/kg, which is within safe limits.
Period: Overall Study
Arm/Group | Human Secretin
Started | 12
Completed | 11
Not Completed | 1
Not completed — Uncooperative/unreliable | 1

BASELINE CHARACTERISTICS:
Groups:
- Human Secretin: Human Secretin : Dose Escalation
Arm/Group | Human Secretin
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: VAS Score at Baseline, Days 1, 2, 3, 4, 7, 30.
Description: 10 point visual analog scale. 0= no pain. 10= worst possible pain. Days 1, 2, 3 were infusion days that included 5 VAS scores each day.
Time Frame: Baseline, Days 1, 2, 3, 4, 7, 30.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Human Secretin
Number analyzed (Participants) | 12
units on a scale
  Baseline | 5.71 (1.45)
  Day 1 Pre-dose | 6.04 (2.13)
  Day 1 Dose 1 (.05mcg/kg) 100min post dose | 4.92 (2.20)
  Day 1 Dose 2 (.1mcg/kg) 100 min post dose | 4.87 (2.06)
  Day 1 Dose 3 (.2mcg/kg) 100 min post dose | 5.30 (2.19)
  Day 1 Dose 3 (.2mcg/kg) 380 min post dose | 4.64 (2.68)
  Day 2 Pre-dose | 5.33 (2.30)
  Day 2 Dose 1 (.1mcg/kg) 100min post dose | 5.25 (1.88)
  Day 2 Dose 2 (.2mcg/kg) 100min post dose | 5.50 (1.71)
  Day 2 Dose 3 (.4mcg/kg) 100min post dose | 4.67 (2.32)
  Day 2 Dose 3 (.4mcg/kg) 380min post dose | 4.77 (2.60)
  Day 3 Pre-dose | 4.92 (2.36)
  Day 3 Dose 1 (.2mcg/kg) 100min post dose | 4.58 (2.15)
  Day 3 Dose 2 (.4mcg/kg) 100min post dose | 4.33 (2.11)
  Day 3 Dose 3 (.8mcg/kg) 100min post dose | 5.17 (2.44)
  Day 3 Dose 3 (.8mcg/kg) 380min post dose | 4.71 (2.47)
  Day 4 | 4.80 (2.49)
  Day 7 | 5.18 (2.62)
  Day 30 | 4.91 (2.20)
Statistical Analysis 1: Comparison: Human Secretin; Change from baseline to day 4; Test type: Superiority or Other; p = .25, t-test, 2 sided
Statistical Analysis 2: Comparison: Human Secretin; Change from baseline to day 7; Test type: Superiority or Other; p = .19, t-test, 2 sided
Statistical Analysis 3: Comparison: Human Secretin; Change from baseline to Day 30; Test type: Superiority or Other; p = .27, t-test, 2 sided

2. Secondary Outcome: Number of Participants With Serious Adverse Events.
Time Frame: 30 Days
Measure: Number; unit: participants
Arm/Group | Human Secretin
Number analyzed (Participants) | 12
participants | 3

3. Primary Outcome: Opiate Use at Baseline, Days 4 and 30.
Description: Daily opiate use (oral morphine equivalent).
Time Frame: Baseline, Day 4, Day 30.
Measure: Mean (Standard Deviation); unit: mg/day
Arm/Group | Human Secretin
Number analyzed (Participants) | 12
mg/day
  Baseline | 139.6 (90.5)
  Day 4 | 127.0 (99.2)
  Day 30 | 97.2 (80.5)
Statistical Analysis 1: Comparison: Human Secretin; Change from baseline to Day 4; Test type: Superiority or Other; p = .52, t-test, 2 sided
Statistical Analysis 2: Comparison: Human Secretin; Change from baseline to Day 30; Test type: Superiority or Other; p = .34, t-test, 2 sided

4. Primary Outcome: Quality of Life at Baseline, Day 4 and Day 30.
Description: Sf-36 ranges from 0 to 151. Higher scores indicating worse outcomes.
Time Frame: Baseline, Day 4, Day 30.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Human Secretin
Number analyzed (Participants) | 12
units on a scale
  Baseline | 100.92 (5.26)
  Day 4 | 100.9 (6.42)
  Day 30 | 101.45 (5.68)

5. Secondary Outcome: VAS Score at Each Administered Dose.
Description: 10 point scare from 0-10 with higher scores meaning higher levels of pain. VAS score assessed after each dose was summarized over Days 1, 2, and 3.
Time Frame: Days 1, 2, and 3.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Human Secretin
Number analyzed (Participants) | 12
units on a scale
  Pre-dose | 6.04 (2.13)
  .05 mcg/kg | 4.92 (2.2)
  .1 mcg/kg | 5.06 (1.94)
  .2 mcg/kg | 4.92 (2.14)
  .4 mcg/kg | 4.5 (2.18)
  .8 mcg/kg | 5.36 (2.46)

ADVERSE EVENTS:
Groups:
- Human Secretin: Human Secretin : Dose Escalation within participant
Arm/Group | Human Secretin
Serious Adverse Events (participants affected / at risk) | 3/12
Other Adverse Events (participants affected / at risk) | 9/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Human Secretin (N=12)
Central line infection (coagulase negative S. Aureus infection with bacteremia) (Infections and infestations) | 1/1 (1) — Previous Hx central line infections. The SAE was related to a PICC line positioned in the R subclavian vein to provide the patient with TPN required by a Dx of CP related to alcohol abuse. Only subject in study with central line so only one at risk.
Pain, nausea, vomitting (Gastrointestinal disorders) | 1 (1)
epigastrium and right upper quadrant pain (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Human Secretin (N=12)
nausea, mild (Gastrointestinal disorders) | 4
mild flushing, upper body (Vascular disorders) | 6 — Flushing is listed as a side effect in the package insert for human secretin.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No